CLINICAL TRIAL: NCT07145047
Title: Clinical Study on the Application of Oncolytic Virus in Recurrent Glioblastoma
Brief Title: Clinical Study of Oncolytic Virus in Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mianyang Central Hospital (Other)
Responsible Party: Principal Investigator, Liangxue Zhou, Dr., Mianyang Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S20230381-02
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma (GBM)
MeSH Terms: conditions — Glioblastoma | interventions — Oncolytic Virotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oncolytic virus in recurrent glioblastoma (Experimental)
  Interventions: Biological: oncolytic virus

INTERVENTIONS:
Biological: oncolytic virus — Intratumoral injection of oncolytic virus.

SUMMARY:
This clinical trial aims to evaluate whether an oncolytic viral agent can treat recurrent glioblastoma. It will also assess the safety and tolerability of the oncolytic viral agent. The primary question it seeks to answer is: What medical problems do participants experience when injected with the oncolytic viral agent? Researchers will administer the oncolytic viral agent via intratumoral injection to determine its efficacy in treating recurrent glioblastoma.

Participant Procedures:

Receive the initial injection, followed by additional injections every 2-4 weeks for a total of 6 injections.

Undergo physical examinations and tests every 2 to 4 weeks. Record their symptoms, hematological test results, and imaging findings.

ELIGIBILITY:
Inclusion criteria:

1. Patients with recurrent glioblastoma, for whom the standard methods of treatment are considered ineffective by the medical commission.
2. Histologically confirmed recurrent glioblastoma.
3. Magnetic resonance imaging (MRI) showed that the maximum diameter of recurrent lesions is greater than 1.0 cm.
4. Before inclusion of patients in the study, at least one of the following types of therapy was previously performed: 4.1 Time from the last radiotherapy/surgery is more than 28 days; 4.2 Subjects maintained stable or declining for at least 7 days prior to corticosteroid regimen; 4.3 Most recent antitumor therapy must have been completed within the specified time prior to treatment: vincristine 2 weeks, nitrosoureas 4 weeks, bevacizumab 4 weeks, temozolomide 6 weeks.
5. Age >=18 years, <=70 years.
6. Hematological indicators, kidney and liver function are normal.
7. The subjects must agree to the use of an acceptable contraceptive method throughout the study, from the time informed consent is provided to 180 days after receiving treatment.
8. Patient's ability to perform the study procedure and provide written informed consent in accordance with the GCP and local laws.

Exclusion criteria:

1. Incompatibility of patients with the inclusion criteria mentioned above.
2. Participated in other drug clinical trials within 4 weeks
3. Preoperative bleeding susceptibility or use of anticoagulants or any medication that may increase the risk of bleeding.
4. Patients with extracranial metastases.
5. Have poorly controlled clinical diseases, such as liver aminotransferase (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)) or total bilirubin > 2 times the upper normal limit.
6. Female subjects: during pregnancy or lactation.
7. Uncontrolled active infection, unstable or severe concomitant disease of infection. Patients with immunodeficiency, autoimmune diseases, active HBV infection, HCV infection, or active HIV infection.
8. Patients with a history of psychotropic substance abuse who are unable to quit or with mental disorders.
9. Subjects had any active autoimmune disease or a history of autoimmune disease.
10. Has a history of antiviral drug use within 1 week.
11. Subjects are receiving immunosuppressive therapy, or concurrent chemotherapy, or radiation, or biotherapy.
12. There are prohibited items for MRI, such as: pacemakers, epicardial pacemaker wires, infusion pumps, surgical and/or aneurysm clips, shrapnel, metal prostheses, potentially magnetic implants, metal objects in the eye, etc..
13. History of substance abuse or known medical, or psychological, or social conditions, such as alcohol or drug abuse.
14. Allergic, hypersensitive or intolerant to study oncolytic viruses (including any excipients).
15. Vaccination within 30 days prior to administration.
16. Patients who have received gene transfer therapy or treated with any type of oncolytic virus.
17. History of encephalitis, or multiple sclerosis, or other central nervous system (CNS) infections, or primary CNS disease.
18. Male or female patients who refused contraception during the study period and for 6 months after dosing.
19. In the investigator's judgment, there is a serious concomitant disease that endangers the patient's safety or interferes with the patient's ability to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 hours, 2 days, 7 days and 14 days after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Mianyang Central Hospital, Mianyang, Sichuan, China

IPD SHARING:
Plan to Share IPD: No